CLINICAL TRIAL: NCT06242561
Title: Quantification of Dilutional Anemia in the Initial Phase of Sepsis Management: Preliminary Retrospective Study: a Preliminary Retrospective Study
Brief Title: Quantification of Dilutional Anemia in the Initial Phase of Sepsis Management: Preliminary Retrospective Study
Acronym: QUADS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-14Obs-CHRMT
Record Dates: First submitted 2024-01-05; First posted 2024-02-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Sepsis
Keywords: hemoglobin levels
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Data collection from sepsis management — observational study

SUMMARY:
This is a single-center retrospective study conducted at Mercy hospital, aiming to investigate the correlation between changes in hemoglobin (Hb) levels and the volume of vascular refill administered during the first 48 hours.

DETAILED DESCRIPTION:
Vascular refill is central to the initial management of hypotension in sepsis, and is often started even before the patient is admitted to intensive care. Over the past 20 years, we have moved from ultraliberal fluid resuscitation to restrictive resuscitation. Indeed, in the early 2000s, the implementation of an early and aggressive hemodynamic optimization strategy, including liberal vascular filling, improved the survival of critically ill patients, and ushered in the era of the Surviving Sepsis Campaign. However, studies have shown increased morbidity and mortality associated with a positive fluid balance. Restrictive approaches to fluid resuscitation and/or deressuscitation were then tested. While these approaches failed to demonstrate any benefit in terms of mortality, they did have the merit of demonstrating their feasibility and good tolerability, albeit with a little-explored pathophysiology. Little is known about the problem of dilutional anemia in the acute phase of septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Patients with septic shock, admitted to Mercy hospital between November 1, 2022 and July 31, 2023, with Noradrenaline administration for at least 6 hours and at least 2 hemoglobin measurements during the first 48 hours of resuscitation.

Exclusion Criteria:

* patients with acute bleeding or blood transfusion before or during the first 48 hours of resuscitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Septic patients
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Total volume of fluids administered during the first 48 hours of ICU stay | 48 hours from ICU admission
  Total volume of fluids (ml)

SECONDARY OUTCOMES:
Haemoglobinemia | 48 hours from ICU admission
  Haemoglobinemia (g/dl)
Type of fluids administered during the first 48 hours of ICU stay | 48 hours from ICU admission
  resuscitation, nutrition, maintenance // crystalloids, colloids, dextrose, sodium bicarbonate
Volume of fluids administered before admission in ICU (ml) | at ICU admission
  Volume of fluids (ml)
In hospital mortality | at hospital discharge : an average of 15 days
  rate
Length of hospital stay | at hospital discharge : an average of 15 days
  Length of hospital stay (days)

CONTACTS AND LOCATIONS:
Overall Officials: Damien BARRAUD, MD, Principal Investigator — CHR Metz Thionville Hopital Mercy
Locations (1):
- CHR Metz-Thionville/Hopital Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No
According to the French law and the French Data Protection Authority (CNIL), we won't be able to publicly share individual participant data, but we plan to share their conclusions through peer-reviewed publications and conferences.